CLINICAL TRIAL: NCT00890045
Title: A Comparison Between the HeRO® Graft and Conventional Arteriovenous Grafts in Hemodialysis Patients
Brief Title: Hemodialysis Reliable Outflow (HeRO) Vascular Access Patency Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merit Medical Systems, Inc. (Industry)
Collaborators: CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-0004
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis
Keywords: Vascular access hemodialysis; ePTFE graft; Graft-eligible; Long-term vascular access for hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control graft (Active Comparator): Conventional ePTFE hemodialysis graft
  Interventions: Device: Conventional ePTFE hemodialysis graft
- HeRO Vascular Access Device (Experimental): HeRO Vascular Access Device
  Interventions: Device: HeRO Vascular Access Device

INTERVENTIONS:
Device: HeRO Vascular Access Device — HeRO Vascular Access Device
  Arms: HeRO Vascular Access Device
Device: Conventional ePTFE hemodialysis graft — Conventional ePTFE hemodialysis graft
  Arms: Control graft

SUMMARY:
Compare the HeRO Vascular Access Device to a conventional ePTFE graft.

DETAILED DESCRIPTION:
The purpose of this study is to compare the HeRO Vascular Access Device to a conventional ePTFE graft. It is hypothesized that HeRO patency will be comparable to the conventional ePTFE graft control.

ELIGIBILITY:
Inclusion Criteria:

1. 22 years of age or older.
2. Male or non-pregnant female.
3. Life expectancy 2 years.
4. End-stage renal disease requiring an arm vascular prosthesis for dialysis access.
5. Ability to understand and provide written informed consent.
6. Willing and able to cooperate with follow-up examinations.
7. Subject's upper arm can be used for implant (Note: The GVAS device must be implanted in the upper arm only, but the Control group graft can be implanted in the upper or lower arm location.).
8. Able to follow a daily aspirin and/or other oral anticoagulation/antiplatelet regimen.

Exclusion Criteria:

1. Potential graft target artery less than 3 mm in diameter determined by any suitable preoperative measure.
2. Documented history of drug abuse within six months.
3. "Planned" concomitant surgical procedure or previous major surgery within 30 days, excluding vascular access related procedures.
4. Currently being treated with another investigational device or drug.
5. Known bleeding diathesis or hypercoagulable state.
6. Peripheral white blood cell count 1500/mm3 (1.5 K/mm3) or platelet counts 50,000/mm3 (50 K/mm3).
7. Degenerative connective tissue disease, e.g., Marfan's and Ehlers Danlos Syndrome. Subjects with Lupus Erythematosus may be included.
8. Subjects with known or suspected concomitant bacterial, fungal, viral, or parasitic infection. Subjects with Hepatitis B may be included. Subjects who are HIV + with CD4 count of <200 are excluded.
9. Severe underlying co-morbidity or immediate life-threatening condition.
10. Subjects with any condition which, in the opinion of the investigator, could preclude evaluation of response or completion of follow-up or affect subject safety.
11. Subjects who are candidates for autologous fistulas.
12. Subjects with scheduled renal transplant within the next 12 months.

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2004-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Glickman, MD, Principal Investigator — Sentara Heart Hospital, Norfolk, VA
Locations (11):
- United States (11):
  - St. Vincent's Medical Center, Los Angeles, California
  - University of Miami/Cedars Medical Center, Miami, Florida
  - St. Joseph's Hospital, Atlanta, Georgia
  - Southern Illinois Unversity, Springfield, Illinois
  - Holy Cross Hospital, Rockville, Maryland
  - North Memorial Medical Center, Robbinsdale, Minnesota
  - Duke Medical Center, Durham, North Carolina
  - Seton/Brackenridge Hospitals, Austin, Texas
  - Baylor Medical Center/Methodist Hospital, Houston, Texas
  - Baptist Medical Center, San Antonio, Texas
  - Sentara Heart Hospital, Norfolk, Virginia

REFERENCES:
- [Result] Nassar GM, Glickman MH, McLafferty RB, Croston JK, Zarge JI, Katzman HE, Peden EK, Lawson JH, Martinez JM, Thackeray L. A comparison between the HeRO graft and conventional arteriovenous grafts in hemodialysis patients. Semin Dial. 2014 May-Jun;27(3):310-8. doi: 10.1111/sdi.12173. Epub 2014 Jan 15. PMID 24428351

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Graft | HeRO Vascular Access Device
Started | 20 | 52 (Of the 52 subjects randomized to the HeRO Graft, two implants were abandoned.)
Completed | 15 | 42
Not Completed | 5 | 10
Not completed — Death | 0 | 1
Not completed — Did not receive HeRO Graft | 0 | 2
Not completed — Lost to Follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Conventional Arteriovenous ePTFE Graft Recipients
- HeRO Group: HeRO Graft Recipients
- Total: Total of all reporting groups
Arm/Group | Control Group | HeRO Group | Total
Number analyzed (Participants) | 20 | 52 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (13.5) | 62.9 (12.5) | 63.8 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 28 | 38
  Male | 10 | 24 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 24 | 38
  White | 5 | 21 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 7 | 8
Region of Enrollment [Number; unit: participants]
  United States | 20 | 52 | 72
History of Coronary artery disease [Number; unit: participants]
  Yes | 15 | 39 | 54
  No | 5 | 13 | 18
History of Diabetes mellitus [Number; unit: participants]
  Yes | 14 | 34 | 48
  No | 6 | 18 | 24
History of Hypertension [Number; unit: participants]
  Yes | 19 | 49 | 68
  No | 1 | 3 | 4
Access History [Number; unit: participants]
  De Novo Access | 5 | 19 | 24
  Re do Access | 15 | 33 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Primary Patency
Description: Primary patency was defined as the interval of time from access placement until any intervention designed to maintain or reestablish patency, access thrombosis, or the time of measurement of patency.
Time Frame: 6 months, 12 months
Population: The denominator represents the number of subjects who are not lost to follow-up, withdrew or died prior to that visit window close date. Note: Of the 52 subjects randomized to the HeRO Graft, 50 subjects were successfully implanted. Two implants were abandoned.
Measure: Number (95% Confidence Interval); unit: percentage of participants patent
Arm/Group | Control Group | HeRO Group
Number analyzed (Participants) | 19 | 49
percentage of participants patent
  6 Months | 48.2 [25.1 to 68.0] | 47.0 [32.7 to 60.1]
  12 Months: number analyzed (Participants) | 18 | 49
  12 Months | 30.6 [11.8 to 51.9] | 34.8 [21.9 to 48.0]

2. Primary Outcome: Percentage of Patients With Assisted Primary Patency
Description: Assisted primary patency was defined as the interval of time from access placement until access thrombosis or the time of measurement of patency, including intervening manipulations (i.e., surgical or endovascular interventions) designed to maintain the functionality of a patent access.
Time Frame: 6 months, 12 months
Population: The denominator represents the number of subjects who are not lost to follow-up, withdrew or died prior to that visit window close date.
Measure: Number (95% Confidence Interval); unit: percentage of participants patent
Arm/Group | Control Group | HeRO Group
Number analyzed (Participants) | 15 | 36
percentage of participants patent
  6 Months | 88.8 [62.1 to 97.1] | 86.2 [71.7 to 93.6]
  12 Months: number analyzed (Participants) | 13 | 32
  12 Months | 75.2 [46.1 to 90.0] | 79.8 [63.1 to 89.5]

3. Primary Outcome: Percentage of Patients With Secondary Patency
Description: Secondary patency was defined as the interval of time from access placement until access abandonment, thrombosis, or the time of patency measurements including intervening surgical or endovascular interventions designed to reestablish functionality in a thrombosed access.
Time Frame: 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants patent
Arm/Group | Control Group | HeRO Group
Number analyzed (Participants) | 19 | 45
percentage of participants patent
  6 Months | 58.4 [33.8 to 76.7] | 76.7 [61.8 to 86.4]
  12 Months: number analyzed (Participants) | 18 | 44
  12 Months | 58.4 [33.8 to 76.7] | 67.6 [52.0 to 79.1]

4. Primary Outcome: Number of Patients With Serious Device or Implant Procedure-related Adverse Events
Description: Serious adverse events were defined as events that required hospitalization ≥24 hours, prolonged an existing hospitalization, resulted in persistent or significant disability or incapacity, were considered life-threatening, or resulted in death.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Control Group | HeRO Group
Number analyzed (Participants) | 20 | 52
participants
  Bleeding, hemorrhage or hematoma | 0 | 6
  Death | 0 | 1
  Device technical failure | 0 | 1
  Embolism | 0 | 2
  Heart failure | 1 | 0
  Infection (non-BSIe) | 2 | 2
  Other | 2 | 5
  Site pain | 0 | 1
  Trauma to major veins, arteries, nerves | 0 | 1
  Steal syndrome | 1 | 2
  Device/Implant procedure-related Bloodstream Infec | 1 | 3

5. Secondary Outcome: Adequacy of Dialysis
Description: Reported as Mean Kt/V, K= dialyzer clearance of urea, t= dialysis time, V=subject total body water
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kt/V
Arm/Group | Control Group | HeRO Group
Number analyzed (Participants) | 10 | 33
Kt/V | 1.7 (0.4) | 1.6 (0.3)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control Group | HeRO Group
Serious Adverse Events (participants affected / at risk) | 5/20 | 19/52
Other Adverse Events (participants affected / at risk) | 4/20 | 5/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=20) | HeRO Group (N=52)
Bleeding, hemorrhage or hematoma (Blood and lymphatic system disorders) | 0 (0) | 6 (6)
Death (General disorders) | 0 (0) | 1 (1)
Device technical failure (General disorders) | 0 (0) | 1 (2)
Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Heart failure (Cardiac disorders) | 0 (0) | 1 (2)
Infection (non-BSI) (Infections and infestations) | 2 (2) | 2 (2)
Other (General disorders) | 2 (2) | 5 (8)
Site pain (General disorders) | 0 (0) | 1 (1)
Trauma to major veins, arteries, nerves (Nervous system disorders) | 0 (0) | 1 (1)
Steal syndrome (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=20) | HeRO Group (N=52)
Right Atrial Clot (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension with fever (Vascular disorders) | 0 (0) | 1 (1)
non-sustained mild and ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
hypoxia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
hypoxemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
elevated white blood cell count (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
symptomatic central venous stenosis (Vascular disorders) | 4 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to slow enrollment and early termination of the study, a shortcoming of this trial, a final conclusion on equivalency between the HeRO Graft and conventional AV graft could not be firmly established.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No